CLINICAL TRIAL: NCT07216677
Title: A Real-World Study of Interventional Clinical Outcomes in Patients With Open Angle Glaucoma and Other Chronic Eye Diseases
Status: Active, not recruiting | Type: Observational
Sponsor: Interstat LLC (Other)
Responsible Party: Principal Investigator, Tsontcho Ianchulev, Ophthalmologist, Interstat LLC
Other Study IDs: CAN-012
Record Dates: First submitted 2025-10-10; First posted 2025-10-14 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Glaucoma; AMD; Diabetic Retinopathy (DR)
Keywords: Glaucoma AMD
MeSH Terms: conditions — Glaucoma; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post-intervention Observational Group
  Interventions: Other: Chronic Disease Intervention CDI

INTERVENTIONS:
Other: Chronic Disease Intervention CDI — Intervention for the management of a chronic eye disease

SUMMARY:
This is a real world investigation of patient who have undergone treatments for chronic eye conditions such as glaucoma and AMD.

DETAILED DESCRIPTION:
The objective of the study is to understand the real-world outcomes after chronic disease treatments for glaucoma and AMD and to compare to reported clinical study outcomes

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Glaucoma or AMD or Diabetic Retinopathy Recent history of a chronic disease intervention in the prior 6 months

Exclusion Criteria:

Patient who are pregnant lactating younger than 18 years of age unable to execute informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a chronic eye disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2027-10-25 (Estimated); Study Completion 2027-10-25 (Estimated)

PRIMARY OUTCOMES:
Changes in Chronic Disease Interventional outcomes such as Intraocular pressure, best corrected vision and other parameters. | up to 12 months
  Longitudinal change in interventional chronic disease outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Interstat, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No